CLINICAL TRIAL: NCT04060719
Title: Effect of Rifampicin on the Pharmacokinetics of a Single Oral Dose of BI 894416 in Healthy Male Subjects (an Open-label, One-way Crossover Study)
Brief Title: A Study in Healthy Men to Test Whether Rifampicin Influences the Amount of BI 894416 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1371-0005; 2019-000507-33 (EudraCT Number)
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reference (Period 1) - BI 894416 alone (Experimental): Reference (Period 1) followed by Test (Period 2)
  Interventions: Drug: BI 894416
- Test (Period 2) - BI 894416 + Rifampicin (Experimental)
  Interventions: Drug: BI 894416; Drug: Rifampicin

INTERVENTIONS:
Drug: BI 894416 — tablet
Drug: Rifampicin — tablet
  Arms: Test (Period 2) - BI 894416 + Rifampicin

SUMMARY:
The main objective of this trial is to investigate the effect of rifampicin on the pharmacokinetics of BI 894416.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG) and including the neurological examination) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (unless the subject quit smoking for at least 3 months prior to first planned administration of trial medication)
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes, but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system). Febrile seizures in childhood or adolescence, recovered carpal tunnel syndrome, recovered uncomplicated meningitis, recovered herpes zoster, tension headache, occasional benign tics (e.g. due to stress) or minor par- or dysesthesia (e.g. as a side effect of prior blood withdrawal) do not constitute a history of relevant neurological disorder.
* History of immunological disease except allergy not relevant to the trial (such as mild hay fever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Liver enzymes (ALT, AST, gGT, AP) above upper limit of normal at the screening examination
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* Male subjects with Woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, 2-treatment, 2-period, 1-way crossover trial to compare the test treatment (T) to the reference treatment (R). The treatments were 1 single dose of BI 894416 following 7 days of pretreatment with rifampicin (T) and 1 single dose of BI 894416 given alone (R) with a washout period of at least 10 days between administrations of BI 894416.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 894416 Alone (Reference)/BI 894416 + Rifampicin (Test): In treatment period 1, Day 1, participants were administered one oral single dose of 50 milligram (mg) BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 milliliter (mL) of water) (reference treatment in period 1, Reference). In treatment period 2, from Day -7 to Day -1, participants were administered one film-coated tablet of 600 mg rifampicin with 240 mL of water once daily, followed by one oral single dose of 50 mg BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 mL of water) on Day 1 (test treatment in period 2, Test). There was a washout period of at least 10 days between the administrations of BI 894416.
Period: Period 1
Arm/Group | BI 894416 Alone (Reference)/BI 894416 + Rifampicin (Test)
Started | 16
Completed | 16
Not Completed | 0
Period: Washout Period
Arm/Group | BI 894416 Alone (Reference)/BI 894416 + Rifampicin (Test)
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2
Arm/Group | BI 894416 Alone (Reference)/BI 894416 + Rifampicin (Test)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all participants who were treated with at least 1 dose of trial drug.
Arm/Group | BI 894416 Alone (Reference)/BI 894416 + Rifampicin (Test)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before administration of BI 894416 and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34 and 48 hours after administration of BI 894416.
Population: Pharmacokinetic (PK) parameter analysis set (PKS) included all participants who were treated with at least 1 dose of trial drug and provided at least 1 PK endpoint defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanomole / liter
Groups:
- BI 894416 Alone (Reference, R): In treatment period 1, Day 1, participants were administered one oral single dose of 50 milligram (mg) BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 milliliter (mL) of water) (reference treatment in period 1, Reference).
- BI 894416 + Rifampicin (Test, T): In treatment period 2, from Day -7 to Day -1, participants were administered one film-coated tablet of 600 mg rifampicin with 240 mL of water once daily, followed by one oral single dose of 50 mg BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 mL of water) on Day 1 (test treatment in period 2, Test).
Arm/Group | BI 894416 Alone (Reference, R) | BI 894416 + Rifampicin (Test, T)
Number analyzed (Participants) | 16 | 16
hour * nanomole / liter | 9077.08 (NA) — Geometric Standard Error (gSE) = 1.09 | 951.58 (NA) — Geometric Standard Error (gSE) = 1.09
Statistical Analysis 1: Comparison: BI 894416 Alone (Reference, R) vs BI 894416 + Rifampicin (Test, T); Relative bioavailability; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; Mixed effects model on the logarithmic scale including effects for 'subject' (random) and 'treatment' (fixed); Adjusted Geometric Mean Ratio T/R [%] = 10.48, 90% CI 2-sided [9.74 to 11.28] — Confidence intervals were calculated based on the residual error from the mixed effects model. Ratio is calculated as Test/Reference. Intra-individual geometric coefficient of variation (gCV) = 11.8

2. Primary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax)
Description: Maximum measured concentration of BI 894416 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole / liter
Arm/Group | BI 894416 Alone (Reference, R) | BI 894416 + Rifampicin (Test, T)
Number analyzed (Participants) | 16 | 16
nanomole / liter | 1624.79 (NA) — Geometric Standard Error (gSE) = 1.10 | 487.98 (NA) — Geometric Standard Error (gSE) = 1.10
Statistical Analysis 1: Comparison: BI 894416 Alone (Reference, R) vs BI 894416 + Rifampicin (Test, T); Relative bioavailability; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; Mixed effects model on the logarithmic scale including effects for 'subject' (random) and 'treatment' (fixed); Adjusted Geometric Mean Ratio T/R [%] = 30.03, 90% CI 2-sided [25.76 to 35.02] — Confidence intervals were calculated based on the residual error from the mixed effects model. Ratio is calculated as Test/Reference. Intra-individual geometric coefficient of variation (gCV) = 25.2

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanomole / liter
Groups:
- BI 894416 Alone (Reference, R): In treatment period 1 participants were administered 1 oral single dose of 50 milligram (mg) BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 milliliter (mL) of water) (Reference, R).
- BI 894416 + Rifampicin (Test, T): In treatment period 2 participants were administered 1 oral single dose of 50 milligram (mg) BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 milliliter (mL) of water) following 7 days of pretreatment with 600 mg rifampicin once daily as tablet formulation (1 film-coated tablet of 600 mg administered with 240 mL of water) (Test, T).
Arm/Group | BI 894416 Alone (Reference, R) | BI 894416 + Rifampicin (Test, T)
Number analyzed (Participants) | 16 | 16
hour * nanomole / liter | 9047.51 (NA) — Geometric Standard Error (gSE) = 1.09 | 939.98 (NA) — Geometric Standard Error (gSE) = 1.09
Statistical Analysis 1: Comparison: BI 894416 Alone (Reference, R) vs BI 894416 + Rifampicin (Test, T); Relative bioavailability; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; Mixed effects model on the logarithmic scale including effects for 'subject' (random) and 'treatment' (fixed); Adjusted Geometric Mean Ratio T/R [%] = 10.39, 90% CI 2-sided [9.66 to 11.18] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: BI 894416 (Reference): From treatment with BI 894416 in treatment period 1 until first treatment with rifampicin in treatment period 2, up to 3 days. Rifampicin: From first treatment with rifampicin in treatment period 2 until treatment with BI 894416 in treatment period 2, up to 7 days. BI 894416 + Rifampicin (Test): From treatment with BI 894416 in treatment period 2 until the individual paricipant's end of trial, up to 15 days.
Description: The treated set included all participants who were treated with at least 1 dose of trial drug. The treated set was used for safety analyses.
Groups:
- BI 894416 (Reference): In treatment period 1, Day 1, participants were administered one oral single dose of 50 milligram (mg) BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 milliliter (mL) of water) (reference treatment in period 1, Reference).
- Rifampicin: In treatment period 2, from Day -7 to Day -1, participants were treated with 600 mg rifampicin once daily as tablet formulation (1 film-coated tablet of 600 mg administered with 240 mL of water).
- BI 894416 + Rifampicin (Test): In treatment period 2, from Day -7 to Day -1, participants were administered one film-coated tablet of 600 mg rifampicin with 240 mL of water once daily, followed by one oral single dose of 50 mg BI 894416 as tablet formulation (2 tablets of 25 mg administered in the fasting state with 240 mL of water) on Day 1 (test treatment in period 2, Test).
Arm/Group | BI 894416 (Reference) | Rifampicin | BI 894416 + Rifampicin (Test)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 16/16 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 894416 (Reference) (N=16) | Rifampicin (N=16) | BI 894416 + Rifampicin (Test) (N=16)
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 3
Chromaturia (Renal and urinary disorders) | 0 | 16 | 0
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04060719/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT04060719/SAP_001.pdf